CLINICAL TRIAL: NCT01711346
Title: A Randomized, Controlled, Single-Blind, 2-Period Crossover Study to Assess the Recovery and Lifespan of Radiolabeled Autologous S303 Treated Red Blood Cells
Brief Title: A Study to Assess the Recovery and Lifespan of Radiolabeled Autologous S303 Treated Red Blood Cells
Acronym: S303 RBC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cerus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: CLI 00073
Record Dates: First submitted 2012-10-17; First posted 2012-10-22 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Focus: Assess Post Infusion Viability of S303 RBCs
MeSH Terms: interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- S303 Red Blood Cells (RBCs) (Experimental): Participants will be assigned to S303 Red Blood Cells (RBCs) and then to Conventional, Untreated Red Blood Cells (RBCs).
  Interventions: Biological: S303 Red Blood Cells (RBCs); Biological: Conventional, untreated Red Blood Cells (RBCs)
- Conventional, Untreated Red Blood Cells (RBCs) (Active Comparator): Participants will be assigned to Conventional, Untreated Red Blood Cells (RBCs) and then to S303 Red Blood Cells (RBCs).
  Interventions: Biological: S303 Red Blood Cells (RBCs); Biological: Conventional, untreated Red Blood Cells (RBCs)

INTERVENTIONS:
Biological: S303 Red Blood Cells (RBCs) — Each subject will receive one intravenous infusion of autologous radiolabeled S303 Red Blood Cells (RBCs) in random order. Each infusion will be approximately 10 to 30 mL.
Biological: Conventional, untreated Red Blood Cells (RBCs) — Each subject will receive one intravenous infusion of autologous radiolabeled Conventional, untreated Red Blood Cells (RBCs) in random order. Each infusion will be approximately 10 to 30 mL.

SUMMARY:
The objective of this study is to assess the post-infusion viability of S-303 Red Blood Cells (RBC) by measuring the 24 hour post-infusion recovery and lifespan of autologous RBCs prepared with the S-303 Treatment System for RBC after storage for 35 days in comparison to conventional untreated RBCs stored for 35 days.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years, of either gender
* Normal health status (as determined by the Investigator review of medical history and blood donor physical exam)
* Complete blood count (CBC); including red blood cell (RBC) indices mean cell volume (MCV), mean cell hemoglobin (MCH), mean cell hemoglobin concentration (MCHC), and RBC distribution width(RDW) and serum chemistry values within normal limits (including calcium, bicarbonate, chloride, inorganic phosphate, potassium, sodium, cholesterol, glucose, total protein, triglycerides, lactate dehydrogenase (LDH), alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, blood urea nitrogen (BUN), creatinine). Values outside of normal reference range thought not to be clinically significant may be allowed with a protocol exception.
* Minimum hemoglobin levels of 13 g/dL for female and 14.5 g/dL for male subjects
* Negative blood donor screening test panel for human immunodeficiency virus (HIV), Hepatitis B virus (HBV), Hepatitis C virus (HCV), human T cell leukemic virus (HTLV), Syphilis, and west nile virus (WNV) (if available)
* Female subjects of childbearing potential and male subjects must agree to use a medically acceptable method of contraception throughout the study periods. A barrier method of contraception must be included, regardless of other methods.
* Meet or exceed American Association of Blood Banks (AABB) guidelines for blood donation (with the exception of travel deferrals).
* Signed and dated informed consent form

Exclusion Criteria:

* • Clinically significant acute or chronic disease (as determined by the Investigator)

  * History of RBC autoantibodies/autoimmune hemolytic anemia, RBC allo-antibodies, or autoimmune disease
  * History of congenital red cell disorders including glucose 6 phosphate dehydrogenase (G-6PD) deficiency
  * Serum ferritin <12 ng/mL
  * Positive direct antiglobulin test (DAT) or indirect antiglobulin test (IAT) at study entry
  * Immunosuppressive therapy (e.g., oral or Intravenous (IV) prednisone) within the past 28 days
  * Treatment with any medication known to affect RBC viability
  * Pregnant or nursing female
  * Male subjects or female subjects of childbearing potential not using effective contraception
  * Participation in another clinical study currently or within the past 28 days
  * Prior exposure to S 303 treated RBCs
  * Pre-existing antibody specific to S 303 treated RBCs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-10; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy: 24 hour post-infusion recovery of autologous Red Blood Cells (RBCs) stored for 35 days | 70 Days
  24 hour post-infusion recovery of autologous RBCs stored for 35 days (assessed using the Food and Drug Administration (FDA)) criteria for evaluation of in vivo RBC studies)
Primary Safety: Incidence of antibody specific to S 303 treated Red Blood Cells (RBCs) | 70 days
  Incidence of antibody specific to S 303 treated RBCs

SECONDARY OUTCOMES:
Secondary Safety: Incidence of adverse events | 70 Days
  Incidence of adverse events
Secondary Efficacy Endpoint | 70 days
  Mean lifespan of autologous red blood cells (RBCs)
Secondary Efficacy Endpoint: | 70 days
  Median lifespan (T50) of autologous red blood cells (RBCs)
Secondary Efficacy Endpoint | 70 days
  Area under the curve (AUC) derived from data points collected for the red blood cell (RBC) lifespan

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Cancelas-Perez, MD, PhD, Principal Investigator — Hoxworth Blood Center, Cincinnati, OH; Jerome L Gottschall, MD, Principal Investigator — BloodCenter of Wisconsin, Milwaukee, WI
Locations (2):
- United States (2):
  - Hoxworth Blood Center, Cincinnati, Ohio
  - BloodCenter of Wisconsin Inc., Milwaukee, Wisconsin